CLINICAL TRIAL: NCT00736099
Title: A 78 Week Open Label Extension to Trials Assessing the Safety and Efficacy of BI 1356 (5 mg) as Monotherapy or in Combination With Other Antidiabetic Medications in Type 2 Diabetic Patients.
Brief Title: Safety and Efficacy of Linagliptin (BI 1356) as Monotherapy or in Combination in Type 2 DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1218.40; 2008-000750-13 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

ARMS (2):
- linagliptin 5 mg (Experimental): open label
  Interventions: Drug: linagliptine 5 mg
- linagliptin 5 mg and pioglitazone 30 mg (Experimental): open label
  Interventions: Drug: linagliptine 5 mg and pioglitazone 30 mg

INTERVENTIONS:
Drug: linagliptine 5 mg — safety and efficacy of linagliptine 5 mg open label
  Arms: linagliptin 5 mg
Drug: linagliptine 5 mg and pioglitazone 30 mg — efficacy and safety of the combination linagliptine and pioglitazone
  Arms: linagliptin 5 mg and pioglitazone 30 mg

SUMMARY:
The objective of the current study is to investigate the safety and tolerability of BI 1356 (5 mg / once daily) given for 78 weeks in different modalities of treatment.

The treatment modalities are determined by the treatment in the blinded trial in which every patient was included previously as BI 1356 in monotherapy (patients in 1218.16 trial), BI 1356 in combination with pioglitazone (patients in 1218.15 trial), BI 1356 added to metformin background (patients in 1218.17 trial) or BI 1356 added to a background therapy of metformin in combination with a sulphonylurea (patients in 1218.18 study)

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent in accordance with the GCP and local legislation.
2. Patients completing the entire treatment period as a double blind trial whether or not they have been treated with rescue medication.

Exclusion criteria:

1. Patients who meet one or more of the withdrawal criteria of the treatment period of the previous trial.
2. Pre-menopausal women (last menstruation =< 1 year prior to signing informed consent) who:

   * are nursing or pregnant,
   * or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, true sexual abstinence (when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of birth control) and vasectomised partners. No exception will be made.
3. Alcohol abuse within the 3 months prior to informed consent that would interfere with trial participation.
4. Drug abuse which, in the opinion of the investigator, would interfere with trial participation.
5. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the trial medication.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2122 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (232):
- United States (13):
  - 1218.40.10003 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1218.40.10014 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 1218.40.10001 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1218.40.10021 Boehringer Ingelheim Investigational Site, Northglenn, Colorado
  - 1218.40.10010 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1218.40.10011 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.40.10016 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1218.40.10002 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.40.10004 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1218.40.10005 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.40.10018 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.40.10007 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.40.10009 Boehringer Ingelheim Investigational Site, Federal Way, Washington
- Argentina (4):
  - 1218.40.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.40.54010 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.40.54011 Boehringer Ingelheim Investigational Site, Mendoza
  - 1218.40.54015 Boehringer Ingelheim Investigational Site, Parque Velez Sarfield
- Austria (2):
  - 1218.40.43001 Boehringer Ingelheim Investigational Site, Graz
  - 1218.40.43005 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (7):
  - 1218.40.32005 Boehringer Ingelheim Investigational Site, Bruges
  - 1218.40.32007 Boehringer Ingelheim Investigational Site, Brussels
  - 1218.40.32006 Boehringer Ingelheim Investigational Site, Edegem
  - 1218.40.32004 Boehringer Ingelheim Investigational Site, Genk
  - 1218.40.32003 Boehringer Ingelheim Investigational Site, Ghent
  - 1218.40.32002 Boehringer Ingelheim Investigational Site, Huy
  - 1218.40.32001 Boehringer Ingelheim Investigational Site, Liège
- Canada (13):
  - 1218.40.01005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.40.01010 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.40.01003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.40.01011 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.40.01006 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1218.40.01009 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.40.01002 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1218.40.01012 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1218.40.01008 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.40.20005 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1218.40.01001 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.40.01004 Boehringer Ingelheim Investigational Site, Montague, Prince Edward Island
  - 1218.40.01007 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (13):
  - 1218.40.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.40.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.40.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.40.86013 Boehringer Ingelheim Investigational Site, Chengdu
  - 1218.40.86009 Boehringer Ingelheim Investigational Site, Dalian
  - 1218.40.86011 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1218.40.86014 Boehringer Ingelheim Investigational Site, Haerbin
  - 1218.40.86008 Boehringer Ingelheim Investigational Site, Qingdao
  - 1218.40.86015 Boehringer Ingelheim Investigational Site, Shanghai
  - 1218.40.86010 Boehringer Ingelheim Investigational Site, Shenyang
  - 1218.40.86007 Boehringer Ingelheim Investigational Site, Wuhan
  - 1218.40.86012 Boehringer Ingelheim Investigational Site, Wuhan
  - 1218.40.86006 Boehringer Ingelheim Investigational Site, Xi'an
- Croatia (2):
  - 1218.40.38605 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1218.40.38604 Boehringer Ingelheim Investigational Site, Slavonski Brod
- Czechia (6):
  - 1218.40.42004 Boehringer Ingelheim Investigational Site, Brno
  - 1218.40.42007 Boehringer Ingelheim Investigational Site, Brno
  - 1218.40.42009 Boehringer Ingelheim Investigational Site, Brno
  - 1218.40.42006 Boehringer Ingelheim Investigational Site, Břeclav
  - 1218.40.42008 Boehringer Ingelheim Investigational Site, Hodonín
  - 1218.40.42003 Boehringer Ingelheim Investigational Site, Olomouc
- Finland (5):
  - 1218.40.35806 Boehringer Ingelheim Investigational Site, Helsinki
  - 1218.40.35801 Boehringer Ingelheim Investigational Site, Kuopio
  - 1218.40.35803 Boehringer Ingelheim Investigational Site, Oulu
  - 1218.40.35805 Boehringer Ingelheim Investigational Site, Seinäjoki
  - 1218.40.35802 Boehringer Ingelheim Investigational Site, Turku
- Germany (8):
  - 1218.40.49028 Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - 1218.40.49022 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.40.49024 Boehringer Ingelheim Investigational Site, Bosenheim
  - 1218.40.49020 Boehringer Ingelheim Investigational Site, Dresden
  - 1218.40.49101 Boehringer Ingelheim Investigational Site, Mainz
  - 1218.40.49003 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.40.49007 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1218.40.49014 Boehringer Ingelheim Investigational Site, Saarbrücken
- Greece (7):
  - 1218.40.30004 Boehringer Ingelheim Investigational Site, Athens
  - 1218.40.30007 Boehringer Ingelheim Investigational Site, Athens
  - 1218.40.30013 Boehringer Ingelheim Investigational Site, Athens
  - 1218.40.30003 Boehringer Ingelheim Investigational Site, Nikaia
  - 1218.40.30011 Boehringer Ingelheim Investigational Site, Piraeus
  - 1218.40.30006 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1218.40.30016 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hungary (6):
  - 1218.40.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.40.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.40.36006 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.40.36008 Boehringer Ingelheim Investigational Site, Debrecen
  - 1218.40.36005 Boehringer Ingelheim Investigational Site, Győr
  - 1218.40.36002 Boehringer Ingelheim Investigational Site, Szombathely
- India (14):
  - 1218.40.91010 Boehringer Ingelheim Investigational Site, Andhra Pradesh
  - 1218.40.91002 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.40.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.40.91012 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.40.91014 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.40.91009 Boehringer Ingelheim Investigational Site, Hyderabad, Andra Pradesh
  - 1218.40.91006 Boehringer Ingelheim Investigational Site, Jaipur
  - 1218.40.91001 Boehringer Ingelheim Investigational Site, Kerala
  - 1218.40.91011 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.40.91008 Boehringer Ingelheim Investigational Site, Mangalore
  - 1218.40.91007 Boehringer Ingelheim Investigational Site, Manipal
  - 1218.40.91004 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.40.91003 Boehringer Ingelheim Investigational Site, Nashik
  - 1218.40.91013 Boehringer Ingelheim Investigational Site, Uttar Pradesh
- Israel (7):
  - 1218.40.97274 Boehringer Ingelheim Investigational Site, Afula
  - 1218.40.97273 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.40.97275 Boehringer Ingelheim Investigational Site, Holon
  - 1218.40.97271 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1218.40.97272 Boehringer Ingelheim Investigational Site, Nahariya
  - 1218.40.97276 Boehringer Ingelheim Investigational Site, Safed
  - 1218.40.97278 Boehringer Ingelheim Investigational Site, Tel Aviv
- Italy (4):
  - 1218.40.39008 Boehringer Ingelheim Investigational Site, Genova
  - 1218.40.39002 Boehringer Ingelheim Investigational Site, Milan
  - 1218.40.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1218.40.39006 Boehringer Ingelheim Investigational Site, Roma
- Japan (5):
  - 1218.40.81001 Boehringer Ingelheim Investigational Site, Amagasaki, Hyogo
  - 1218.40.81005 Boehringer Ingelheim Investigational Site, Koganei, Tokyo
  - 1218.40.81002 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.40.81004 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1218.40.81003 Boehringer Ingelheim Investigational Site, Suita, Osaka,
- Malaysia (6):
  - 1218.40.60007 Boehringer Ingelheim Investigational Site, George Town
  - 1218.40.60003 Boehringer Ingelheim Investigational Site, Kelantan
  - 1218.40.60001 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1218.40.60002 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1218.40.60004 Boehringer Ingelheim Investigational Site, Perak
  - 1218.40.60005 Boehringer Ingelheim Investigational Site, Perak
- Mexico (10):
  - 1218.40.52007 Boehringer Ingelheim Investigational Site, Aguascalientes, Ags.
  - 1218.40.52010 Boehringer Ingelheim Investigational Site, Col.Americana, Guadalajara, Jalisco
  - 1218.40.52008 Boehringer Ingelheim Investigational Site, Colonia Tlalpan, Mexico
  - 1218.40.52006 Boehringer Ingelheim Investigational Site, Faccionamiento Lomas de Campestre,AGUASCAL
  - 1218.40.52009 Boehringer Ingelheim Investigational Site, León
  - 1218.40.52002 Boehringer Ingelheim Investigational Site, México
  - 1218.40.52004 Boehringer Ingelheim Investigational Site, México
  - 1218.40.52005 Boehringer Ingelheim Investigational Site, México
  - 1218.40.52003 Boehringer Ingelheim Investigational Site, Monterrey
  - 1218.40.52001 Boehringer Ingelheim Investigational Site, Monterrey N.L.
- Netherlands (5):
  - 1218.40.31006 Boehringer Ingelheim Investigational Site, Deurne
  - 1218.40.31001 Boehringer Ingelheim Investigational Site, Ewijk
  - 1218.40.31010 Boehringer Ingelheim Investigational Site, Losser
  - 1218.40.31008 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 1218.40.31002 Boehringer Ingelheim Investigational Site, Wildervank
- New Zealand (5):
  - 1218.40.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 1218.40.64003 Boehringer Ingelheim Investigational Site, Dunedin
  - 1218.40.64002 Boehringer Ingelheim Investigational Site, Otahuhu
  - 1218.40.64001 Boehringer Ingelheim Investigational Site, Tauranga
  - 1218.40.64005 Boehringer Ingelheim Investigational Site, Wellington
- Philippines (5):
  - 1218.40.63003 Boehringer Ingelheim Investigational Site, Greenhills, San Juan
  - 1218.40.63005 Boehringer Ingelheim Investigational Site, Manila
  - 1218.40.63002 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.40.63001 Boehringer Ingelheim Investigational Site, Pasig
  - 1218.40.63004 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (3):
  - 1218.40.48603 Boehringer Ingelheim Investigational Site, Lublin
  - 1218.40.48601 Boehringer Ingelheim Investigational Site, Warsaw
  - 1218.40.48604 Boehringer Ingelheim Investigational Site, Zabrze
- Romania (7):
  - 1218.40.40504 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1218.40.40604 Boehringer Ingelheim Investigational Site, Brasov
  - 1218.40.40501 Boehringer Ingelheim Investigational Site, Bucharest
  - 1218.40.40502 Boehringer Ingelheim Investigational Site, Bucharest
  - 1218.40.40603 Boehringer Ingelheim Investigational Site, Galati
  - 1218.40.40503 Boehringer Ingelheim Investigational Site, Sibiu
  - 1218.40.40505 Boehringer Ingelheim Investigational Site, Târgu Mureş
- Russia (11):
  - 1218.40.70014 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 1218.40.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.40.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.40.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.40.70012 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.40.70005 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1218.40.70006 Boehringer Ingelheim Investigational Site, Perm
  - 1218.40.70013 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1218.40.70015 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.40.70016 Boehringer Ingelheim Investigational Site, Samara
  - 1218.40.70004 Boehringer Ingelheim Investigational Site, Tomsk
- Slovakia (6):
  - 1218.40.42103 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1218.40.42102 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.40.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.40.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.40.42101 Boehringer Ingelheim Investigational Site, Nové Mesto
  - 1218.40.42106 Boehringer Ingelheim Investigational Site, Šamorín
- South Korea (11):
  - 1218.40.82002 Boehringer Ingelheim Investigational Site, Busan
  - 1218.40.82011 Boehringer Ingelheim Investigational Site, Daegu
  - 1218.40.82008 Boehringer Ingelheim Investigational Site, Incheon
  - 1218.40.82010 Boehringer Ingelheim Investigational Site, Jeonju
  - 1218.40.82004 Boehringer Ingelheim Investigational Site, Pusan
  - 1218.40.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.40.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.40.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.40.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.40.82009 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.40.82003 Boehringer Ingelheim Investigational Site, Suwon
- Spain (12):
  - 1218.40.34002 Boehringer Ingelheim Investigational Site, Badalona
  - 1218.40.34011 Boehringer Ingelheim Investigational Site, Badia Del Vallés
  - 1218.40.34012 Boehringer Ingelheim Investigational Site, Borges Del Camp
  - 1218.40.34013 Boehringer Ingelheim Investigational Site, Centelles
  - 1218.40.34007 Boehringer Ingelheim Investigational Site, Granada
  - 1218.40.34008 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1218.40.34009 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1218.40.34004 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.40.34006 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.40.34010 Boehringer Ingelheim Investigational Site, Sant Adrià Del Besós (Barcelona)
  - 1218.40.34005 Boehringer Ingelheim Investigational Site, Seville
  - 1218.40.34014 Boehringer Ingelheim Investigational Site, Vic (Barcelona)
- Sweden (4):
  - 1218.40.46013 Boehringer Ingelheim Investigational Site, Härnösand
  - 1218.40.46001 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.40.46012 Boehringer Ingelheim Investigational Site, Uddevalla
  - 1218.40.46004 Boehringer Ingelheim Investigational Site, Uppsala
- Taiwan (8):
  - 1218.40.88605 Boehringer Ingelheim Investigational Site, Changhua
  - 1218.40.88604 Boehringer Ingelheim Investigational Site, Taichung
  - 1218.40.88606 Boehringer Ingelheim Investigational Site, Tainan
  - 1218.40.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.40.88602 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.40.88603 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.40.88607 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.40.88608 Boehringer Ingelheim Investigational Site, Taoyuan District
- Thailand (2):
  - 1218.40.66001 Boehringer Ingelheim Investigational Site, Bangkok
  - 1218.40.66002 Boehringer Ingelheim Investigational Site, Khon Kaen
- Ukraine (12):
  - 1218.40.38011 Boehringer Ingelheim Investigational Site, Dnipro
  - 1218.40.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.40.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.40.38010 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.40.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.40.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.40.38008 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.40.38009 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.40.38012 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.40.38003 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.40.38006 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1218.40.38007 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (9):
  - 1218.40.44005 Boehringer Ingelheim Investigational Site, Ashford
  - 1218.40.44004 Boehringer Ingelheim Investigational Site, Baillieston, Glasgow
  - 1218.40.44001 Boehringer Ingelheim Investigational Site, Bath
  - 1218.40.44003 Boehringer Ingelheim Investigational Site, Burbage
  - 1218.40.44010 Boehringer Ingelheim Investigational Site, Bury Saint Edmonds
  - 1218.40.44009 Boehringer Ingelheim Investigational Site, Cardiff
  - 1218.40.44002 Boehringer Ingelheim Investigational Site, Penarth
  - 1218.40.44006 Boehringer Ingelheim Investigational Site, Reading
  - 1218.40.44007 Boehringer Ingelheim Investigational Site, Waterloo, Liverpool

RESULTS

PARTICIPANT FLOW:
Groups:
- Old Lina: Patients pre-treated with linagliptin (BI 1356)
- New Lina: Patients pre-treated with placebo
Period: Overall Study
Arm/Group | Old Lina | New Lina
Started | 1532 (Number who started treatment.) | 589 (Number who started treatment.)
Completed | 1349 (Number who completed treatment.) | 531 (Number who completed treatment.)
Not Completed | 183 | 58
Not completed — Adverse Event | 61 | 18
Not completed — Protocol Violation | 10 | 4
Not completed — Lost to Follow-up | 12 | 5
Not completed — Withdrawal by Subject | 42 | 13
Not completed — Lack of Efficacy | 15 | 8
Not completed — Other reason | 43 | 10

BASELINE CHARACTERISTICS:
Groups:
- Old Lina: Patients pre-treated with linagliptin
- Total: Total of all reporting groups
Arm/Group | Old Lina | New Lina | Total
Number analyzed (Participants) | 1532 | 589 | 2121
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.8) | 56.7 (10.0) | 57.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 743 | 279 | 1022
  Male | 789 | 310 | 1099
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.86 (4.82) | 29.18 (4.91) | 28.95 (4.85)
Baseline weight [Mean (Standard Deviation); unit: kg] | 78.7 (16.9) | 80.1 (16.9) | 79.1 (16.9)
Baseline Glycosylated haemoglobin (HbA1c) at baseline [Mean (Standard Deviation); unit: percent] | 7.38 (0.90) | 7.87 (1.04) | 7.51 (0.97)
Fasting plasma glucose (FPG) at baseline [Mean (Standard Deviation); unit: mg/dL] | 151.59 (35.32) | 164.31 (37.36) | 155.12 (36.34)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Patients With Adverse Events (AEs)
Description: This includes any AEs detected during routine physical examination and electrocardiogram (ECG) procedures.
Time Frame: 78 weeks
Population: Treated Set: all screened patients who were documented to have taken at lease 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1532 | 589
Participants
  Patients with any AEs | 1253 | 465
  Patients with severe AEs | 57 | 23
  Patients with withdrawal due to AEs (from AE page) | 57 | 16

2. Primary Outcome: Frequency of Patients With Investigator-defined Hypoglycaemic Adverse Events
Time Frame: 78 weeks
Population: Treated Set: all screened patients who were documented to have taken at lease 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1532 | 589
Participants | 209 | 86

3. Primary Outcome: Frequency of Patients With Significant Adverse Events Based on Standardised MedDRA Query (SMQ)
Description: As significant adverse events are considered: renal Aes (SMQ 'acute renal failure'), hypersensitivity reactions ('anaphylactic reactions' and 'angioedema'), hepatic Aes ('hepatitis, non-infectious', 'hepatic failure, fibrosis, cirrhosis and other liver damage-related conditions', 'liver-related investigations, signs and symptoms', 'cholestasis and jaundice of hepatic origin'), severe cutaneous adverse reactions ('severe cutaneous adverse reaction'), pancreatitis ('acute pancreatitis', 'chronic pancreatitis'').
Time Frame: 78 weeks
Population: Treated Set: all screened patients who were documented to have taken at lease 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1532 | 589
Participants
  Renal AEs | 20 | 10
  Hypersensitivity reactions | 7 | 3
  Hepatic AEs | 21 | 5
  Severe cutaneous adverse reactions | 0 | 0
  Pancreatitis | 4 | 0

4. Primary Outcome: Frequency of Patients With Adjudication of Cardiac and Cerebrovascular Events
Description: Patients reported with cardiac and cerebrovascular events qualified for adjudication by the Clinical Event Committee (CEC)
Time Frame: 78 weeks
Population: Treated Set: all screened patients who were documented to have taken at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1532 | 589
participants | 82 | 37

5. Primary Outcome: Number of Patients With Abnormalities in Vital Signs
Description: Vital sign abnormalities (any abnormalities found during PE or ECG are reported with adverse events)
Time Frame: 78 weeks
Population: Treated Set: all screened patients who were documented to have taken at lease 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1532 | 589
Participants | 0 | 0

6. Primary Outcome: Number of Patients With Abnormalities in Haematology: Eosinophils
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than or equal to 10%.
Time Frame: 78 weeks
Population: Treated Set with values for Eosinophils
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1512 | 579
participants | 91 | 33

7. Primary Outcome: Number of Patients With Abnormalities in Haematology: Haemoglobin
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than or equal to 11.5 g/dL for male and as a value less than or equal to 9.5 g/dL for female patients.
Time Frame: 78 weeks
Population: Treated Set with values for Haemoglobin
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1513 | 579
Participants | 63 | 31

8. Primary Outcome: Number of Patients With Abnormalities in Haematology: Haematocrit
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than or equal to 32%.
Time Frame: 78 weeks
Population: Treated Set with values for Haematocrit
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1513 | 579
Participants | 48 | 22

9. Primary Outcome: Number of Patients With Abnormalities in Haematology: Red Blood Cell Count
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 3 * 10^12/L.
Time Frame: 78 weeks
Population: Treated Set with values for Red blood cell count
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1513 | 579
Participants | 31 | 13

10. Primary Outcome: Number of Patients With Abnormalities in Haematology: White Blood Cell Count
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 3 * 10^9/L (decrease) or a value greater than 20.1 * 10^9/L (increase).
Time Frame: 78 weeks
Population: Treated Set with values for White blood cell count
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1513 | 579
Participants
  Decrease | 30 | 10
  Increase | 1 | 1

11. Primary Outcome: Number of Patients With Abnormalities in Haematology: Platelets
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as value less than or equal to 75 * 10^9/L (decrease) or a value greater than or equal to 700 * 10^9/L (increase).
Time Frame: 78 weeks
Population: Treated Set with values for Platelets
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1513 | 579
Participants
  Decrease | 5 | 0
  Increase | 0 | 0

12. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Potassium
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 3 mmol/L (decrease) or a value greater than 5.8 mmol/L (increase).
Time Frame: 78 weeks
Population: Treated Set with values for Potassium
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants
  Decrease | 3 | 0
  Increase | 135 | 50

13. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Uric Acid
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than 11 mg/dL for male and as a value greater than 10 mg/dL for female patients.
Time Frame: 78 weeks
Population: Treated Set with values for Uric acid
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
Participants | 124 | 48

14. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Triglycerides
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than 300 mg/dL.
Time Frame: 78 weeks
Population: Treated Set with values for Triglycerides
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
Participants | 329 | 101

15. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Amylase
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than 1.5 times the upper limit of normal (ULN).
Time Frame: 78 weeks
Population: Treated Set with values for Amylase
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
Participants | 92 | 35

16. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: γ-Glutamyl-transferase (GGT)
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than or equal to 3 times the ULN.
Time Frame: 78 weeks
Population: Treated Set with values for GGT
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
Participants | 54 | 14

17. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Creatinine
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than or equal to 1.5 mg/dL.
Time Frame: 78 weeks
Population: Treated Set with values for Creatinine
Measure: Number; unit: Participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
Participants | 52 | 18

18. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Creatinine Kinase
Description: as for outcome 16
Time Frame: 78 weeks
Population: Treated Set with values for Creatinine kinase
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants | 49 | 6

19. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Phosphate
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 0.7 mmol/L (decrease) or a value greater than 1.7 mmol/L (increase).
Time Frame: 78 weeks
Population: Treated Set with values for Phosphate
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants
  Decrease | 11 | 8
  Increase | 38 | 11

20. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Calcium
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 1.8 mmol/L (decrease) or a value greater than 3 mmol/L (increase).
Time Frame: 78 weeks
Population: Treated Set with values for Calcium
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants
  Decrease | 36 | 12
  Increase | 4 | 0

21. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Sodium
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 130 mmol/L (decrease) or a value greater than 160 mmol/L (increase).
Time Frame: 78 weeks
Population: Treated Set with values for Sodium
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants
  Decrease | 16 | 3
  Increase | 13 | 8

22. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Alanine Transaminase (ALT)
Description: as for outcome 16
Time Frame: 78 weeks
Population: Treated Set with values for ALT
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1511 | 578
participants | 22 | 5

23. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Aspartate Transaminase (AST)
Description: as for outcome 16
Time Frame: 78 weeks
Population: Treated Set with values for AST
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1511 | 578
participants | 19 | 3

24. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Glucose
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 54 mg/dL.
Time Frame: 78 weeks
Population: Treated Set with values for Glucose
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants | 7 | 1

25. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Bilirubin
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than or equal to 2 mg/dL.
Time Frame: 78 weeks
Population: Treated Set with values for Bilirubin
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants | 6 | 3

26. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Alkaline Phosphatase (AP)
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value greater than or equal to 2 times the ULN.
Time Frame: 78 weeks
Population: Treated Set with values for AP
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants | 7 | 0

27. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Albumin
Description: For this laboratory parameter, a possibly clinically significant abnormality is defined as a value less than 2.5 g/dL.
Time Frame: 78 weeks
Population: Treated Set with values for Albumin
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants | 3 | 1

28. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Lactate Dehydrogenase (LDH)
Description: as for outcome 16
Time Frame: 78 weeks
Population: Treated Set with values for LDH
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1511 | 577
participants | 1 | 0

29. Secondary Outcome: Change in HbA1c From Baseline to Week 6
Time Frame: Baseline and week 6
Population: Treated Set with values for HbA1c at baseline and week 6. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1401 | 530
percent | -0.02 (0.47) | -0.46 (0.51)

30. Secondary Outcome: Change in HbA1c From Baseline to Week 18
Time Frame: Baseline and week 18
Population: Treated Set with values for HbA1c at baseline and week 18. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1302 | 510
percent | 0.03 (0.63) | -0.63 (0.72)

31. Secondary Outcome: Change in HbA1c From Baseline to Week 30
Time Frame: Baseline and week 30
Population: Treated Set with values for HbA1c at baseline and week 30. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1183 | 469
percent | 0.06 (0.71) | -0.60 (0.78)

32. Secondary Outcome: Change in HbA1c From Baseline to Week 42
Time Frame: Baseline and week 42
Population: Treated Set with values for HbA1c at baseline and week 42. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1091 | 440
percent | 0.13 (0.65) | -0.53 (0.78)

33. Secondary Outcome: Change in HbA1c From Baseline to Week 54
Time Frame: Baseline and week 54
Population: Treated Set with values for HbA1c at baseline and week 54. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1008 | 417
percent | 0.19 (0.70) | -0.45 (0.81)

34. Secondary Outcome: Change in HbA1c From Baseline to Week 66
Time Frame: Baseline and week 66
Population: Treated Set with values for HbA1c at baseline and week 66. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 949 | 399
percent | 0.14 (0.73) | -0.44 (0.85)

35. Secondary Outcome: Change in HbA1c From Baseline to Week 78
Time Frame: Baseline and week 78
Population: Treated Set with values for HbA1c at baseline and week 78. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 904 | 373
percent | 0.12 (0.76) | -0.49 (0.85)

36. Secondary Outcome: Number of Patients With HbA1c<7.0% Over Time
Time Frame: 78 weeks
Population: Treated Set with values for HbA1c at baseline and week 78. Values after rescue therapy are set to missing.
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 904 | 373
participants | 382 | 172

37. Secondary Outcome: Number of Patients With HbA1c<6.5% Over Time
Time Frame: 78 weeks
Population: Treated Set with values for HbA1c at baseline and week 78. Values after rescue therapy are set to missing.
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 904 | 373
participants | 139 | 74

38. Secondary Outcome: Number of Patients With Lowered HbA1c by at Least 0.5% Over Time
Time Frame: 78 weeks
Population: Treated Set with values for HbA1c at baseline and week 78. Values after rescue therapy are set to missing.
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 904 | 373
participants | 155 | 175

39. Secondary Outcome: Change in FPG From Baseline to Week 6
Time Frame: Baseline and week 6
Population: Treated Set with values for FPG at baseline and at week 6. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1413 | 531
mg/dL | 1.21 (30.54) | -15.17 (30.84)

40. Secondary Outcome: Change in FPG From Baseline to Week 18
Time Frame: Baseline and week 18
Population: Treated Set with values for FPG at baseline and at week 18. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1270 | 499
mg/dL | 2.13 (31.47) | -13.92 (33.54)

41. Secondary Outcome: Change in FPG From Baseline to Week 30
Time Frame: Baseline and week 30
Population: Treated Set with values for FPG at baseline and at week 30. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1166 | 466
mg/dL | 1.52 (31.84) | -16.17 (33.00)

42. Secondary Outcome: Change in FPG From Baseline to Week 42
Time Frame: Baseline and week 42
Population: Treated Set with values for FPG at baseline and at week 42. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1073 | 437
mg/dL | 2.97 (31.07) | -11.87 (31.27)

43. Secondary Outcome: Change in FPG From Baseline to Week 54
Time Frame: Baseline and week 54
Population: Treated Set with values for FPG at baseline and at week 54. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1004 | 416
mg/dL | 3.44 (30.52) | -12.62 (30.96)

44. Secondary Outcome: Change in FPG From Baseline to Week 66
Time Frame: Baseline and week 66
Population: Treated Set with values for FPG at baseline and at week 66. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 955 | 398
mg/dL | 0.88 (31.96) | -12.87 (30.16)

45. Secondary Outcome: Change in FPG From Baseline to Week 78
Time Frame: Baseline and week 78
Population: Treated Set with values for FPG at baseline and at week 78. Values after rescue therapy are set to missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 904 | 366
mg/dL | 1.90 (34.11) | -13.64 (31.67)

46. Primary Outcome: Number of Patients With Abnormalities in Clinical Chemistry: Cholesterol
Description: as for outcome 14
Time Frame: 78 weeks
Population: Treated Set with values for Cholesterol
Measure: Number; unit: participants
Arm/Group | Old Lina | New Lina
Number analyzed (Participants) | 1514 | 579
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 78 weeks
Arm/Group | Old Lina | New Lina
Serious Adverse Events (participants affected / at risk) | 158/1532 | 52/589
Other Adverse Events (participants affected / at risk) | 784/1532 | 285/589
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Old Lina (N=1532) | New Lina (N=589)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 4
Angina pectoris (Cardiac disorders) | 4 | 3
Angina unstable (Cardiac disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 6
Myocardial ischaemia (Cardiac disorders) | 2 | 2
Right ventricular failure (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Dolichocolon (Congenital, familial and genetic disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Peritoneal cyst (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Chest discomfort (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 5 | 2
Generalised oedema (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Polyp (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Vaccination site hypersensitivity (General disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Polyarteritis nodosa (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Amoebic dysentery (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter intestinal infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 0
Chikungunya virus infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Snake bite (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 4 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Intra-uterine contraceptive device removal (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Old Lina (N=1532) | New Lina (N=589)
Nasopharyngitis (Infections and infestations) | 164 | 62
Upper respiratory tract infection (Infections and infestations) | 122 | 54
Urinary tract infection (Infections and infestations) | 74 | 33
Hyperglycaemia (Metabolism and nutrition disorders) | 376 | 121
Hypoglycaemia (Metabolism and nutrition disorders) | 200 | 85
Back pain (Musculoskeletal and connective tissue disorders) | 69 | 31
Hypertension (Vascular disorders) | 67 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.